CLINICAL TRIAL: NCT03397420
Title: Effect of Family-centered Model of HIV Care (FAM-CARE) on Viral Suppression and Retention in Care of HIV-positive Children in Swaziland
Brief Title: Family-centered HIV Care, Viral Suppression and Retention in HIV-positive Children, Swaziland
Acronym: FAM-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Ministry of Health, Swaziland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EG0168
Record Dates: First submitted 2018-01-02; First posted 2018-01-12 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAM-CARE (Experimental): Two facility "clusters" (one hospital and one health center, with their filter clinics) will be randomized to initiate the FAM-CARE program (where all HIV-positive family members are seen together as a unit and receive care together) with viral load monitoring
  Interventions: Other: FAM-CARE
- Control Standard of Care (Active Comparator): Two "clusters" (one hospital and one health center, with their filter clinics) will be control standard-of care (usual practice) sites. Standard HIV care and treatment services, (drug resupply, clinical assessments etc.), including viral load monitoring, will be provided to adults and children in separate adult and pediatric clinics, even though they many be from the same family.
  Interventions: Other: FAM-CARE

INTERVENTIONS:
Other: FAM-CARE — Family-centered care, where all HIV-positive family members are seen together as a unit and receive HIV care and treatment services together, for HIV-positive children and their caregivers

SUMMARY:
The study will evaluate the effect of implementing a family-centered care (FAM-CARE) program (where all HIV-positive family members are seen together as a unit and receive care together) on viral suppression and retention in HIV-positive children <15 years through enrollment of a prospective cohort of 660 HIV-positive children and their caregivers at sites that were randomized to either implement the family-care program (intervention sites) or continue the current standard of care (control sites).

DETAILED DESCRIPTION:
The proposed study will evaluate the effect of implementing a FAM-CARE program on viral suppression and retention in children through enrollment of a prospective cohort of HIV-positive children and their caregivers at sites implementing the FAM-CARE program and control sites continuing the current standard of care. The study will be conducted in four "clusters" of facilities (2 hospitals and 2 health centers and their filter clinics) in the Hhohho region of Swaziland. Two facility "clusters" (one hospital and one health center, with their filter clinics) will be randomized to initiate the FAM-CARE program with viral load monitoring and two "clusters" (one hospital and one health center, with their filter clinics) will be control standard-of care sites. A prospective cohort of HIV-positive children and their caregivers will be followed in the FAM-CARE program sites and control sites. Each child will be followed for 18 months following enrollment. The primary objective is to evaluate the effect of the FAM-CARE program on the rates of viral suppression and retention in care, comparing rates of viral suppression and retention in children enrolled in FAM-CARE versus control sites. The study will also evaluate factors associated with viral suppression and retention (including family demographic characteristics), and conduct qualitative interviews to assess the acceptability of the FAM-CARE program by caregivers and health care providers in the intervention sites.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive child aged <15 years receiving HIV care at the study facility.

Exclusion Criteria:

* At least one family member residing in the household is also HIV-positive and is receiving services at the study facility

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 742 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of HIV-positive children on ART virally suppressed | 18 months after study enrollment.
  Proportion of HIV-positive children on ART with viral suppression (defined as HIV RNA copies/mL below the level of assay detection) and the proportion with HIV RNA <1,000 copies/mL at 18 months after enrollment
Proportion of HIV-positive on ART virally unsuppressed | 18 months after study enrollment.
  Proportion of HIV-positive children on ART with HIV RNA >1000 copies/mL 18 months after enrollment into the study.

SECONDARY OUTCOMES:
Proportion HIV-positive children on ART virally suppressed (<1,000 copies/mL of HIV RNA) at 6 and 12 months after study enrollment | 6 and 12 months after study enrollment
  Proportion of HIV-positive children on ART with viral suppression (defined as HIV RNA copies/mL below the level of assay detection) and HIV RNA >1000 copies/mL
Factors associated with HIV viral suppression | 18 months after study enrollment
  Individual and family factors associated with viral suppression.
Loss to follow-up | 18 months after study enrollment
  Loss to follow-up (not seen in clinical care >3 months)
ART initiation | 18 months after study enrollment
  ART initiation in HIV-positive children not on ART at study entry
Acceptability of the FAM-CARE program based on individual interview responses | 18 months after study enrollment
  Acceptability of the FAM-CARE program to caregivers and health care provider as measured from responses on individual interviews using a structured questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Caspian Chouraya, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Nobuble Mthethwa, MD, Principal Investigator — Ministry of Health, Swaziland; Lynne Mofenson, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- Mbabane, Mbabane, Eswatini

IPD SHARING:
Plan to Share IPD: Yes
All collected IPDs
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Six months after study publication
Access Criteria: Datasets will be available for download upon request from Population Council/USAID website

REFERENCES:
- [Derived] Ashburn K, Chouraya C, Khumalo P, Mpango L, Mthethwa N, Machekano R, Guay L, Mofenson LM. A randomized controlled trial evaluating the effects of a family-centered HIV care model on viral suppression and retention in care of HIV-positive children in Eswatini. PLoS One. 2021 Aug 24;16(8):e0256256. doi: 10.1371/journal.pone.0256256. eCollection 2021. PMID 34428241